CLINICAL TRIAL: NCT01058824
Title: Relative Bioavailability Study Of Two Lincomycin Hydrochloride Hard Gelatinous Capsule 500 Mg Formulations, In Healthy Volunteers Using Formulations (Frademicina®) Manufactured By Pfizer Laboratories Ltd
Brief Title: Relative Bioavailability Study Of Two Lincomycin Hydrochloride Hard Gelatinous Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: B1601001; STPh40/09
Record Dates: First submitted 2010-01-27; First posted 2010-01-29 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Bacterial Infections
Keywords: Bioequivalence; Lincomycin Hydrocloride
MeSH Terms: conditions — Bacterial Infections | interventions — Lincomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lincomycin - Active Comparative - Hard Gelatin Capsule (Active Comparator)
  Interventions: Drug: Lincomycin
- Lincomycin - Study Drug - Hard Gelatin Capsule (Experimental)
  Interventions: Drug: Lincomycin

INTERVENTIONS:
Drug: Lincomycin — Single Dose Hard Gelatin Capsule - oral - 500 mg
  Other Names: Lincomycin Hydrocloride
  Arms: Lincomycin - Active Comparative - Hard Gelatin Capsule
Drug: Lincomycin — Single Dose Hard Gelatin Capsule - oral - 500 mg
  Other Names: Lincomycin Hydrocloride
  Arms: Lincomycin - Study Drug - Hard Gelatin Capsule

SUMMARY:
To assess the relative bioavailability of two different batches of Frademicina® drug product, containing 500 mg lincomycin hydrocloride, manufactured by Pfizer Laboratories Ltd. The formulations' comparative bioavailability after oral administration will be assessed based on the statistical comparisons of the relevant pharmacokinetic parameters, obtained from the drug concentrations in the blood. The lincomycin hydrocloride concentration will be measured by a proper and validated analytical method.

ELIGIBILITY:
Inclusion Criteria:

* Men.
* Women who are not pregnant nor nursing.
* Age between 18 and 50 years-old.
* Body mass index ≥ 19 and ≤ 28,5.
* Good health conditions or with no significant diseases, under judgement of the legally qualified professional, according to the rules defined in the Protocol, and based on the following assessments: clinical history, pressure and pulse measurements, physical and psychological examination, ECG and complementary laboratorial tests.
* Ability to understand the nature and the objective of the trial, including the risks and adverse effects and, agreeing to cooperate with the investigator and to act according to the requirements of the whole assay, which will be confirmed through the signature of the Free Informed Consent.

Exclusion Criteria:

* Known hypersensitivity to the study drug (lincomycin hydrocloride) or to compounds chemically related.
* History or presence of hepatic, gastrointestinal diseases or other conditions that may interfere with the absorption, distribution, excretion or metabolism process of the drug.
* History of hepatic, renal, pulmonary, gastrointestinal, epileptic, hematological or psychiatric condition; of hypo or hypertension from any etiology that require pharmacological treatment; history or had myocardial infarction, angina and/or cardiac insufficiency.
* Electrocardiographic findings non-recommended for the enrollment in the trial, by investigator's criteria.
* Results of the laboratory tests are out of the normal range, according to the standards of this protocol, unless they are considered clinically irrelevant by the investigator.
* He/She is a smoker.
* Drinks more than 05 cups of coffee or tea per day.
* History of alcohol or drug abuse.
* Use of regular medication within 02 weeks prior to the beginning of the treatment and to the assessment date; or use of any medication within a week, except for contraceptive medications.
* Hospitalization for any reason within 08 weeks prior to the beginning of the first treatment period of this trial and to the assessment date.
* Treatment within 03 months prior to the trial with any drug with known toxic potential on primary organs.
* Enrollment to any experimental trial or use of any experimental drug within 06 months prior to the beginning of this trial and to the assessment date.
* Donation or loss of 450 mL or more of blood within 03 months that precede the trial or donation higher than 1500 mL within the 12 months between the beginning of the clinical trial and the assessment date.
* Consumption of inducing and/or inhibiting enzymatic drugs (CYP450 - hepatic), toxic to organ or with long half-life period, within 04 weeks prior to the beginning of the trial.
* Consumption of alcohol within 48 hours preceding the enrollment to the trial and during the clinical trial.
* Consumption of food and beverages that contained grapefruit up to 07 days prior to each trial period.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
AUC [0-t]Area under the curve of concentration vs. time, from time 0 (zero) up to the time of the last observed concentration above the limit of quantification, calculated by the trapezium rules. | 1 week
Cmax Maximum reached concentration, based on the experimental data, obtained directly from the curve concentration vs. time; | 1 week

SECONDARY OUTCOMES:
AUC [0-¥]Area under the curve of drug concentration versus time, from time 0 (zero) extrapolated to the infinite, calculated as AUC [0-¥] = AUC [0-t] + Ct/Ke, in which Ct is the last concentration determined above the limit of | 1 week
quantification. | 1 week
Ke Terminal First Order Elimination Constant, estimated by the angular coefficient of the linear regression, calculated by the Least Square Method, from the natural logarithms of concentration vs. time to the last four values of concentration (or at | 1 week
least three) above the limit of quantification. | 1 week
T½ Half-life time, calculated as ln (2) / Ke. | 1 week
Adverse events and vital signs. | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Campinas, São Paulo, Brazil

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1601001&StudyName=Relative%20Bioavailability%20Study%20Of%20Two%20Lincomycin%20Hydrochloride%20Hard%20Gelatinous%20Capsule